CLINICAL TRIAL: NCT05778110
Title: Multiomic Analysis of Traumatic Brain Injury and Hypertension Intracranial Hemorrhage Lesion Tissue
Acronym: MOSS-THINK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Junfeng Feng, Director of Brain Injury Center, RenJi Hospital
Other Study IDs: LY2023-017-B
Record Dates: First submitted 2023-02-05; First posted 2023-03-21 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Brain Injury Traumatic Severe; Intracranial Hemorrhage, Hypertensive
Keywords: Traumatic brain injury; Hypertensive intracranial hemorrhage; Multiomic analysis; Biomarker; Molecular mechanism
MeSH Terms: conditions — Intracranial Hemorrhage, Hypertensive; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TBI: Patients with traumatic brain injury.
  Interventions: Other: Type of disease
- ICH: Patients with hypertensive intracranial hemorrhage.
  Interventions: Other: Type of disease

INTERVENTIONS:
Other: Type of disease — Different types of pathogen: brain injury by trauma or intracranial hemorrhage due to hypertension.

SUMMARY:
The goal of this experimental observation study is to figure out differently expressed biomarkers in lesion tissues in traumatic brain injury or hypertension intracranial hemorrhage patients. The main questions it aims to answer is:

* Which RNA, protein and metabolites are differently expressed in lesion tissues?
* What molecular mechanism is participated in TBI or ICH? Participants will be treated by emergency operation, and their lesion tissues will be collected during the operation.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 and <65
2. Within 12 hours after brain injury
3. GCS ≥3 and ≤8
4. Closed brain injury with frontotemporal contusion or basal ganglia intracranial hemorrhage
5. Need emergency intracranial hematoma evacuating operation
6. Patient's agents are informed and consent the research

Exclusion Criteria:

1. With TBI, stroke, ICH or intracranial tumor history
2. Death within 24 hours
3. Immunosuppression state
4. Severe organ dysfunction
5. Complicated infective disease
6. Pregnant

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with severe traumatic brain injury or hypertensive intracranial hemorrhage.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
RNA biomarkers in TBI or ICH patients' lesion tissues assessed by transcriptome bioinformatic analysis | Immediately after collecting tissues
  Patients' lesion tissue will be collected during hematoma evacuation. Then these tissues will be immediately prepared to be detected through transcriptome sequencing. The results of transcriptome sequencing will be further analyzed by bioinformatic analysis to reveal different RNA expressions in lesion tissues of severe TBI and ICH patients as the potential biomarkers.
Protein biomarkers in TBI or ICH patients' lesion tissues assessed by proteomic bioinformatic analysis | Immediately after collecting tissues
  Patients' lesion tissue will be collected during hematoma evacuation. Then these tissues will be immediately prepared to be detected through proteomics mass spectrometry. The results of proteomic will be further analyzed by bioinformatic analysis to reveal different protein expressions in lesion tissues of severe TBI and ICH patients as the potential biomarkers.
Metabolite biomarkers in TBI or ICH patients' lesion tissues assessed by metabolomic bioinformatic analysis | Immediately after collecting tissues
  Patients' lesion tissue will be collected during hematoma evacuation. Then these tissues will be immediately prepared to be detected through metabolomic mass spectrometry. The results of metabolomic will be further analyzed by bioinformatic analysis to reveal different metabolite expressions in lesion tissues of severe TBI and ICH patients as the potential biomarkers.

CONTACTS AND LOCATIONS:
Locations (1):
- Brain Injury Center, Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No